CLINICAL TRIAL: NCT06557954
Title: Cervical Cytology DNA Methylation for Cervical Cancer Screening: A Real Word Study
Brief Title: Cervical Cytology DNA Methylation for Cervical Cancer Screening
Status: Not yet recruiting | Type: Observational
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: METHY5
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cervical Cancer; DNA Methylation; Cytology; Human Papillomavirus Infection; Cervical Intraepithelial Neoplasia; Cancer Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: human PAX1 and JAM3 gene methylation assays (PAX1m/JAM3m) — PAX1m/JAM3m, with or without HPV testing and cytological pathology for cervical cancer screening
  Other Names: HPV testing; cytological pathology

SUMMARY:
Cervical cancer represents one of the foremost causes of cancer-related morbidity and mortality among women worldwide. Given the current limitations, such as the low specificity of human papillomavirus (HPV) testing and the relatively low sensitivity of cytological examinations, there is a pressing need for a novel, non-invasive, safe, and precise screening method. This study aims to undertake a multicentre, real-world investigation, incorporating at least 10 sub-centres and enrolling 30,000 participants. Histopathological examination results will serve as the 'gold standard' for evaluating the screening efficacy of human PAX1 and JAM3 gene methylation assays (PAX1m/JAM3m), HPV testing, and cytological examinations. Furthermore, the study seeks to elucidate the relationship between DNA methylation levels and persistent HPV infection, while also assessing the applicability of PAX1m/JAM3m across diverse clinical settings. By focusing on alterations in DNA methylation levels within cervical exfoliated cells as the primary research trajectory, this study aspires to furnish novel insights and theoretical foundations for the prevention and management of cervical cancer, targeting PAX1m/JAM3m. The ultimate objective is to facilitate the clinical implementation of an enhanced cervical cancer screening protocol, thereby addressing the deficiencies of current screening methodologies, achieving greater precision in cervical cancer screening, and effectively reducing the incidence of cervical cancer while mitigating the risks of overdiagnosis and overtreatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* With uterine cervix intact
* Given consents to participate the study
* With detailed follow-up outcomes

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women asking for cervical cancer screening in hospital situation or in community situationg
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with histopathological diagnosis of grade 2 cervical intraepithelial neoplasia (CIN) or worse (CIN2+) | 1 year
  Including CIN2, CIN3, adenocarcinoma in situ and invasive cervical carcinoma
Number of participants with histopathological diagnosis of grade 3 cervical intraepithelial neoplasia (CIN) or worse (CIN3+) | 1 year
  Including CIN3, adenocarcinoma in situ and invasive cervical carcinoma

SECONDARY OUTCOMES:
Number of participants with histopathological diagnosis of invasive cervical carcinoma | 1 year
  Including invasive cervical carcinoma of various subtypes

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No